CLINICAL TRIAL: NCT04347395
Title: Prevention of Respiratory Infections in Older Patients During and After Hospitalisation: A Randomised Controlled Trial
Brief Title: Respiratory Infection in Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015/3138
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pneumonia; Respiratory Infection; Dysphagia
Keywords: clinical trial; pneumonia; vaccination; geriatric; respiratory infection; dysphagia
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Control Group (No Intervention): Current best practice for prevention of HAP
- Group 2: Intervention (Experimental): Respiratory Bundle Intervention
  Interventions: Procedure: Respiratory Bundle & Prevention

INTERVENTIONS:
Procedure: Respiratory Bundle & Prevention — The respiratory care bundle intervention comprised of: bed tilt, swallow screen, mouth wash and vaccinations. The bed tilt was a 30-degree whole bed-up positioning both day and night throughout the hospital stay and is shown in Figure 1. Swallow screen was undertaken within 48 hours of admission. Chlorhexidine mouth wash was prescribed initially four times daily. The protocol was amended to twice daily chlorhexidine mouth wash in August 2017 due to poor compliance with four times daily administration. Mouthwash administration was monitored in the intervention group only and deemed non-compliant if missed more than 3 times during the admission. Pneumococcal and influenza vaccination was offered at discharge or within 2-4 weeks post discharge, at no charge to the patient. Post discharge advice was to use pillows in bed to minimize the time the patient laid flat and to avoid lying down for an hour after meals.
  Arms: Group 2: Intervention

SUMMARY:
This randomized controlled trial in older hospitalized patients found that a respiratory care bundle intervention did not significantly reduce the incidence of respiratory infections compared to usual care for the index admission. However, time to next admission for respiratory infection was significantly longer with the intervention compared to usual care.

Aim: To evaluate whether a respiratory care bundle, compared to usual care, reduces respiratory infections during and after hospitalization.

Methods: In this open-label, single-centre randomized controlled trial, we recruited patients >65 years of age and admitted <72 hours for non-respiratory conditions to a novel respiratory care bundle intervention (whole bed tilt, swallow screen, chlorhexidine mouth wash, and pneumococcal and influenza vaccinations) or usual care. Participants were followed up for 12 months. The primary endpoint was the development of respiratory infection during the index admission. The secondary endpoint was the time to next admission for respiratory infection.

DETAILED DESCRIPTION:
Background:

Hospital-acquired infections impact patient recovery and increase risk of deterioration. Pneumonia is the second commonest cause of death in Singapore accounting for 19% of deaths in 2014. Hospital acquired pneumonia (HAP) or nosociomal pneumonia refers to any pneumonia contracted by a patient in a hospital at least 48-72 hours after admission and is usually caused by a bacterial infection, rather than a virus. It is the most prevalent hospital-acquired infection, and has the highest mortality among the hospital-acquired infections (20-50%) . Local audit data has shown that around 60% of deaths in hospitalised older patients are due to pneumonia, of which a significant proportion are due to HAP or health care associated pneumonia (HCAP).

A meta-analysis of respiratory studies has shown low numbers of studies evaluating novel antimicrobial agents for hospital-acquired pneumonia (15.9%) suggesting further research or novel approaches are needed. The prevalence of nosociomal pneumonia in a European study was 13.9%. Pneumonia acquired during periods of hospitalisation has a high morbidity, mortality and increased hospital length of stay (LOS). Audit of the 2014 data from the Geriatric Mortality meetings has shown all cause pneumonia (community acquired pneumonia (CAP) and HAP) is 55%. Currently this data is being analysed to calculate the proportion of deaths attributable to HAP vs CAP.

The pathophysiology of pneumonia in the elderly is primarily due to aspiration pneumonia (ASP). ASP comprises predominantly two pathological conditions: airspace infiltration with bacterial pathogens and dysphagia-associated aspiration. The primary route of infection is believed to be through microaspiration of organisms that have colonised the oropharynx and gastrointestinal tract. Hospitalised patients become colonised with microorganisms from the hospital environment within 48 hours and severity of respiratory infection is related to the number and virulence of these microorganisms as well as the hosts immune response.

Swallowing difficulties, poor oral hygiene and reduced immune response are inherent in the older population contributing to an increased risk of HAP. In addition, older patients have an increased risk of aspiration of gastric contents due to a laxity of lower oesphageal sphincter, an anatomical sphincter that relies on diaphragmatic function. Many older patients locally are fed via naso-gastric tube and the presence of a naso-gastric tube increases the risk of aspiration pneumonia occuring during hospitalisation. Supine positioning also predisposes to micro aspiration from the oropharynx and stomach with many patients placed routinelyin a supine position to undertake their basic care needs. Positioning in the semi recumbant position has been shown to reduce microaspiration with elevations of 30-45 degrees by improving supraglottic drainage.

Patients cared for in intensive care units have been shown to benefit from a targeted bundle of care that reduced ventilator associated pneumonia (VAP) and it is therefore likely that these principles could be extended to benefit older patients. The VAP bundle includes head up tilt (30 degrees), gastric acid suppression and good oral hygiene. In this study, gastric acid suppression will not be used routinely as some studies have suggested that the use of proton pump inhibitors may increase the risk of HAP. Research has shown reduced pneumonia rates and hospital re-admissions after the implementation of good oral care methods and a local quality improvement project (Bright Smiles) has been shown to improve the quality of oral care in older patients. Assessment of swallowing function at an early stage within the hospital admission offers the opportunity to identify earlier those patients with swallowing difficulties and intervene to reduce the likelihood of aspiration.

In a Spanish prospective multicenter case-control study of patients with HCAP or CAP more than 50% were due to streptococcus pneumoniae and the presence of multiple co-morbidities were associated with HCAP. In older patients with multiple co-morbidities there is poor uptake of vaccination and therefore the utilization of a vaccination programme for these patients proposes to reduce the likelihood of re-admission due to HCAP or HAP and aims to impact the hospital re-admission rates in geriatric patients.

The local data has identified the need for a novel approach to hospital acquired infections and the techniques described have shown benefit in ventilated patients but this study aims to extend the principle of preventing aspiration to a wider population of "at risk" older patients through positioning, swallowing assessment and good oral care.

The study planned is a randomized control trial (intervention arm vs control arm) to compare current best practice with a respiratory bundle of care.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized geriatric patients >65 years age
* likely hospital length of stay >72 hours.

Exclusion Criteria:

* participants < 65 years;
* spinal cord injury;
* pneumonia or chest infection as admission diagnosis;
* active cancer of the respiratory tract;
* pressure ulcer grade 3, grade 4 or unstageable;
* hospital admission likely to be <72 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
In Older Patients (>65 years age) | 9.5months
  To reduce the incidence of HAP

SECONDARY OUTCOMES:
In Older Patients (>65 years age) | 9.5months
  To reduce the 90 day mortality from HAP To reduce the hospital 30 day re-admission rate for Geriatric patients To reduce the 90 day re-admission rate for HCAP in Geriatric patients

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Rosario BH, Shafi H, Yii ACA, Tee LY, Ang ASH, Png GK, Ang WST, Lee YQ, Tan PT, Sahu A, Zhou LF, Zheng YL, Slamat RB, Taha AAM. Evaluation of multi-component interventions for prevention of nosocomial pneumonia in older adults: a randomized, controlled trial. Eur Geriatr Med. 2021 Oct;12(5):1045-1055. doi: 10.1007/s41999-021-00506-3. Epub 2021 Jun 3. PMID 34081314